CLINICAL TRIAL: NCT03101670
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Study to Assess the Efficacy and Safety of Filgotinib Administered for 16 Weeks to Subjects With Moderately to Severely Active Psoriatic Arthritis
Brief Title: A Study to Assess Efficacy and Safety of Filgotinib in Active Psoriatic Arthritis
Acronym: EQUATOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-224
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- filgotinib (Experimental)
  Interventions: Drug: filgotinib
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: filgotinib — one filgotinib oral tablet q.d.
  Arms: filgotinib
Drug: Placebo Oral Tablet — one placebo oral tablet q.d.
  Arms: placebo

SUMMARY:
This is a multicenter, Phase 2, double-blind, placebo-controlled study in subjects with moderately to severely active Psoriatic Arthritis (PsA) who have an inadequate response or are intolerant to conventional disease-modifying therapy. A total of approximately 124 subjects will be randomized to one of 2 treatment arms in a 1:1 ratio: oral filgotinib tablets q.d. or matching placebo tablets q.d. The Screening visit will occur within 28 days before study drug administration. At Day 1 (Baseline), eligible subjects will be randomized to treatment for a duration of 16 weeks. The study is concluded with a Follow-up period lasting until 4 weeks after the last dose. Consequently, each subject will stay in the study for a maximum of 24 weeks (from Screening visit to Follow-up visit).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects who are ≥18 years of age, on the day of signing informed consent.
* Diagnosis of psoriatic arthritis meeting Classification Criteria for Psoriatic Arthritis (CASPAR)
* Have active psoriatic arthritis defined as ≥5 swollen joints (from a 66 swollen joint count [SJC]) and ≥5 tender joints (from a 68 tender joint count [TJC]) at Screening and Baseline (measurable dactylitis of a digit counts as a single swollen joint and if tender, then also a single tender joint).
* Have had a history of documented plaque psoriasis or currently active plaque psoriasis
* If using cDMARD therapy, subjects must have been on it for 12 weeks prior to screening, with a stable dose (including stable route of administration) for at least 4 weeks prior to baseline.
* If using non-drug therapies (including physical therapies), thse should be kept sable during screening
* Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use highly effective methods of contraception as described in the protocol

Key Exclusion Criteria:

* Use of JAK inhibitors, investigational or approved, at any time, including filgotinib;
* Prior use of more than one TNF inhibitor, at any time.
* Use of oral steroids at a dose >10 mg/day of prednisone or prednisone equivalent or at a dose that hasn't been stable for at least 4 weeks prior to Baseline;
* Any therapy by intra-articular injections (e.g. corticosteroid, hyaluronate) within 4 weeks prior to screening;
* Use of more than 1 NSAID or cyclooxygenase-2 (COX-2) inhibitor.
* Have undergone surgical treatment for psoriatic arthritis including synovectomy and arthroplasty in more than 3 joints and/or within the last 12 weeks prior to screening
* Presence of very poor functional status or unable to perform self-care.
* Administration of a live or attenuated vaccine within 12 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who have reached ACR20 response as compared to placebo | Week 16
  To assess the effect of filogotinib on PsA as assessed by ACR20 in PsA patients

SECONDARY OUTCOMES:
Assessment of minimal disease activity (MDA) in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on MDA in PsA patients
Percentage of subjects who have reached ACR50 response as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsA as assessed by ACR50 in PsA patients
Percentage of subjects who have reached ACR70 response as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsA as assessed by ACR70 in PsA patients
Percentage of subjects achieving DAS28(CRP) score as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsA as assessed by DAS28 (CRP) in PsA patients
Percentage of subjects achieving SDAI response as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsA as assessed by SDAI response in PsA patients
Percentage of subjects achieving CDAI response as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on PsA as assessed by CDAI response in PsA patients
Percentage of subjects achieving EULAR response as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsA as assessed by EULAR response in PsA patients
Assessment of psoriatic arthritis response criteria (PsARC) as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on PsARC in PsA patients
Assessment of physician's and patient's global assessment of disease activity as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on physician's and patient's global assessment of disease activity in PsA patients
Assessment of patient's global assessment of PsA pain intensity in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on on PsA pain intensity in PsA patients
Assessment of joints for tenderness (68) and swelling (66) in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on joint tenderness and swelling in PsA patients
Assessment of CRP in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filogotinib on CRP in PsA patients
Psoriasis as assessed by PASI in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on PASI in PsA patients
Psoriasis as assessed by PASI50 in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on PASI50 in PsA patients
Psoriasis as assessed by PASI75 in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the affect of filgotinib on PASI75 in PsA patients
Psoriasis as assessed by PASI90 in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the affect of filgotinib on PASI90 in PsA patients
Psoriasis as assessed by PASI100 in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the affect of filgotinib on PASI100 in PsA patients
Physician's and patient's global assessment of psoriasis in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the affect of filgotinib on Physician's and patient's global assessment of psoriasis in PsA patients
Assessment of mNAPSI in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on mNAPSI in PsA patients
Assessment of pruritis NRS in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on NRS in PsA patients
Enthesitis as assessed by SPARCC enthesitis index in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on SPARCC enthesitis index in PsA patients
Dactilytis as assessed by LDI in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on Dactilytis in PsA patients
Physical function as assessed by HAQ-DI in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on physical function in PsA patients
FACIT-Fatigue scale in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on FACIT-Fatigue scale in PsA patients
Assessment of SF-36 in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on SF-36 in PsA patients
Assessment of Psoriatic Arthritis Impact of Disease Questionnaire (PsAID) in filgotinib treated subjects as compared to placebo | At each visit from screening until the final follow up visit (week 20)
  To assess the effect of filgotinib on PsAID in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects in the number of adverse events | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal clinical laboratory evaluations | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal vital signs | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal physical examination | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal ECG | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal radiographic assessment | From screening until the final follow up visit (week 20)
  To evaluation safety and tolerability of filgotinib in PsA patients

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, DPhil, MRCP (UK), Study Director — Galapagos NV
Locations (25):
- ULB Hopital Erasme, Service de Rheumatology, Brussels, Belgium
- Bulgaria (4):
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - UMHAT "SofiaMed", OOD, Block 1, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
- Czechia (2):
  - CCBR Czech, a.s, Pardubice
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Estonia (3):
  - Center for Clinical and Basic Research, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - OÜ Innomedica, Tallinn
- Poland (4):
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól
  - Ai Centrum Medyczne sp. z o.o. sp.k., Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Przychodnia Specjalistyczna, Torun
  - Centrum Medyczne AMED, Warszawa Targowek, Warsaw
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Servicio de Reumatologia, Fuenlabrada
  - Hospital Infanta Luisa, Servicio de Reumatologia, Seville
- Ukraine (9):
  - CI of Healthcare Kharkiv CCH #8 Dept of Rheumatology Kharkiv MA of PGE of MOHU, Ch of Cardiology and Funct Diagnostics, Kharkiv
  - CNI Consultative and Diagnostic Center of Pecherskyi District of Kyiv, Department of Therapy, Kiev
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Unit of Non-coronary HD&Rh, Kiev
  - CH of State Border Service of Ukraine (Military Base 2522) Dept of Therapy, D.Halytskyi Lviv NMU, Ch of Family Medicine & Dermatology, Venereology, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Rheumatology HSEIU UMSA, Ch of Family Medicine and Therapy, Poltava
  - CI of TRC, Ternopil
  - M.I. Pyrogov VRCH Dept of Rheumatology M.I. Pyrogov VNMU, Ch of IM #1, Vinnytsia
  - MCIC MC LLC Health Clinic, Unit of Cardiology and Rheumatology, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Un of Therapy and CRh Dept of Therapy, Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chandran V, Malkov VA, Ito KL, Liu Y, Vestergaard L, Yoon OK, Liu J, Trivedi M, Hertz A, Gladman D. Pharmacodynamic effects of filgotinib treatment driving clinical improvement in patients with active psoriatic arthritis enrolled in the EQUATOR trial. RMD Open. 2023 Nov;9(4):e003550. doi: 10.1136/rmdopen-2023-003550. PMID 37945284
- [Derived] Orbai AM, Ogdie A, Gossec L, Tillett W, Leung YY, Gao J, Trivedi M, Tasset C, Meuleners L, Besuyen R, Hendrikx T, Coates LC. Effect of filgotinib on health-related quality of life in active psoriatic arthritis: a randomized phase 2 trial (EQUATOR). Rheumatology (Oxford). 2020 Jul 1;59(7):1495-1504. doi: 10.1093/rheumatology/kez408. PMID 31624837
- [Derived] Mease P, Coates LC, Helliwell PS, Stanislavchuk M, Rychlewska-Hanczewska A, Dudek A, Abi-Saab W, Tasset C, Meuleners L, Harrison P, Besuyen R, Van der Aa A, Mozaffarian N, Greer JM, Kunder R, Van den Bosch F, Gladman DD. Efficacy and safety of filgotinib, a selective Janus kinase 1 inhibitor, in patients with active psoriatic arthritis (EQUATOR): results from a randomised, placebo-controlled, phase 2 trial. Lancet. 2018 Dec 1;392(10162):2367-2377. doi: 10.1016/S0140-6736(18)32483-8. Epub 2018 Oct 22. PMID 30360969